CLINICAL TRIAL: NCT07276789
Title: A Phase 2, Open-Label, Multicenter Study to Investigate the Efficacy and Safety of a Single Dose of LS301-IT for Fluorescence Intraoperative Molecular Imaging (IMI) for Lung Cancer Resection
Brief Title: Efficacy and Safety of a Single Dose of LS301-IT for Fluorescence Intraoperative Molecular Imaging (IMI) for Patients Undergoing Lung Cancer Resection for Non Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Integro Theranostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS301-IT-B201
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: lung cancer; lung cancer resection; Non Small Cell Lung Cancer Resection; Non-Small Cell Lung Cancer Stage I-II
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: A single-dose, open-label, multicenter, Phase 2 study in patients scheduled to undergo minimally invasive surgery (MIS) for known or suspected lung cancer via thoracoscopy (i.e., VATS or RATS). Single dose IV infusion of 0.1 mg/kg of LS301-IT given up to 4 days before surgery. There will be no stratification by dosing interval, type of minimally invasive surgery, or tumor type.
Masking Description: Pathologist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LS301-IT 1.0 mg/kg (Experimental)
  Interventions: Drug: LS301-IT 0.1 mg/kg

INTERVENTIONS:
Drug: LS301-IT 0.1 mg/kg — Single dose of LS301-IT administed up to 4 days prior to surgery

SUMMARY:
The aim of this Phase 2 study is to investigate the efficacy and safety of a single dose of LS301-IT, a novel fluorescence imaging agent developed by Integro Theranostics (IT), administered by intravenous (IV) infusion in patients undergoing VATS (Video-Assisted Thoracoscopic Surgery) or RATS (Robotic-Assisted Thoracoscopic Surgery) resection of Stage I-II non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
The primary objective of the study is to determine the proportion of subjects that have at least one Clinically Significant Event (CSE) using fluorescence imaging, defined as either the localization of the primary tumor when white light has failed to identify the tumor, the identification of a synchronous or occult pulmonary tumor with fluorescence only, or the identification of an inadequate surgical margin after resection. Secondary objectives include the determination of the sensitivity and positive predictive value (PPV) of LS301 fluorescence imaging in the identification of tumor using histopathology as the gold standard, and the assessment of the safety and tolerability of LS301-IT. Exploratory objectives include the determination of the "Clinical Impact Rate" defined as the proportion of cases when the surgeon changes the scope of the procedure based on LS301 fluorescence imaging, the assessment of the dosing interval prior to surgery, and the standardization of imaging during surgery and surgeon assessment of fluorescence.

ELIGIBILITY:
Inclusion Criteria

* Have a primary diagnosis, or a high clinical suspicion, for cancer in the lung based on CT, biopsy, or other imaging.
* Are scheduled to undergo surgical thoracoscopy and resection of the lung.
* If of childbearing potential, the patient must have a negative serum pregnancy test at screening, on Day 1 prior to LS301-IT administration, as well as using a medically acceptable form of contraception (eg, hormonal birth control, double-barrier method) or abstinence.
* Ability to understand the requirements of the study

Exclusion Criteria:

* Contraindications for surgery or any medical condition that in the opinion of the investigator could jeopardize the safety of the subject
* History of any drug-related hypersensitivity or anaphylactic reactions, including those attributed to indocyanine green (ICG) or other contrast agents.
* Patients with impaired renal function
* History, or presence in the ECG at Screening, of any clinically significant abnormalities including cardiac conduction abnormalities
* History of radiation therapy to the chest
* Total bilirubin level >1.5 times upper limit
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) > 2.5 times the upper limit of normal (ULN)
* Patient is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Clinically Significant Events | On the day of surgery
  To determine the proportion of subjects that have at least one CSE where a CSE is defined as one of 3 possible clinical events:
  a. Identification of primary tumor in situ with fluorescence IMI after non-ID with white light b. Identification of synchronous or occult lung tumors with fluorescence IMI after non-ID with white light c. Identification of tumor margin of resected specimen ex vivo within 10 mm of staple line with fluorescence IMI (both ≤5 mm and ≤10 mm will be assessed)

SECONDARY OUTCOMES:
Sensitivity | day or surgery
  The number of patients that are true positive divided by the number of patients that are true positive + the number of patients that are false positive (True Positive/True Positive + False Negative) of fluorescence IMI using intraoperative surgeon assessment with histopathology as the gold standard
Positive Predictive Value | day of surgery
  Number of patients that are true positive divided by the number of patients that are true positive + false positive (True Positive/(True Positive + False Positive) of fluorescence IMI using intraoperative surgeon assessment with histopathology as the gold standard
Primary tumor identification rate | day of surgery
  Proportion of patients that underwent flourescent imaging where the primary tumor was identified by flourescence
Synchronous or occult tumor identification rate | day of surgery
  Propotion of the total number of synchronous or occult tumors identified by flourescent imaging
Close margin rate | day of surgery
  The proportion of patients with a close margin identified by fluorescent imaging. Close margin is defined as a margin within less than or equal to 5 mm from the staple line and less than or equal to 10 mm from the staple line
Incidence of Adverse Events | within 30 days after dosing
  The proportion of patients reporting at least one adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Robert Honigberg, MD, Study Director — Integro Theranostics
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
As the study is an early stage study, there is no current plan to share the IPD.